CLINICAL TRIAL: NCT03005275
Title: A Comparison of Cost - Effectiveness of Stimulated ICSI and IVM Strategy in PCOS Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam National University (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Director, Vietnam National University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NCKH/CGRH-04-2016
Record Dates: First submitted 2016-12-19; First posted 2016-12-29 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVM (Other): * FSH injection: Day 9, 10 and 11 (can be adjusted 1-3 days before or after to avoid Ultrasound and OPU on holidays). Dose: normally 100 IU/day (maybe 75 - 150 IU/day).
  * Follicle and endometrium can be evaluated: on the day of final injection or one day later.
  * hCG 10.000 IU: one day after the final FSH injection, at 9 p.m. Can be adjusted HCG injection day (± 1-2 days) to avoid Ultrasound and OPU on vacation.
  * OPU: 1,5 day after hCG injection (normally 36-42 hours later).
  * Sperm collection: on OPU day (if mature follicle presents) or 1 day after OPU day.
  * Embryo transfer: 3 days after OPU.
  * Luteal support: progesterone gel (90 mg once daily) intra-vaginally and estradiol (4 mg/day PO, twice daily) initiated on the day of OPU or the day thereafter.
  Interventions: Other: IVM
- ICSI (Other): Daily SC injections with rFSH (minimum starting dose is around 150 IUI) are started on On day 2 or day 3 of the menstrual cycle (Stimulation Day 1) and continue up to and including Stimulation Day 7.
  From Stimulation Day 8 onwards, subjects from ICSI treatment groups will continue with a daily SC dose of rFSH up to the day before GnRH agonist day. The maximum rFSH dose to continue treatment after the first 7 days is 300 IU but the dose could be adjusted when desired.
  As soon as three follicles of 17mm are observed by USS at least, a GnRH agonist (Triptorelin 0.2 mg) will be used for final oocyte maturation at the same day. About 34-36 h thereafter, OPU followed by ICSI is performed. Two days after oocyte pick-up 2 fresh embryos will be transferred.
  Interventions: Other: ICSI

INTERVENTIONS:
Other: IVM — FSH injection: Day 9, 10 and 11 (can be adjusted 1-3 days before or after to avoid Ultrasound and OPU on holidays). Dose: normally 100 IU/day (maybe 75 - 150 IU/day).
  Follicle and endometrium can be evaluated: on the day of final injection or one day later.
  hCG 10.000 IU: one day after the final FSH injection, at 9 p.m. Can be adjusted HCG injection day (± 1-2 days) to avoid Ultrasound and OPU on vacation.
  OPU: 1,5 day after hCG injection (normally 36-42 hours later). Sperm collection: on OPU day (if mature follicle presents) or 1 day after OPU day.
  Embryo transfer: 3 days after OPU. Luteal support: progesterone gel (90 mg once daily) intra-vaginally and estradiol (4 mg/day PO, twice daily) initiated on the day of OPU or the day thereafter.
  Arms: IVM
Other: ICSI — Daily SC injections with rFSH (minimum starting dose is around 150 IUI) are started on On day 2 or day 3 of the menstrual cycle (Stimulation Day 1) and continue up to and including Stimulation Day 7.
  From Stimulation Day 8 onwards, subjects from ICSI treatment groups will continue with a daily SC dose of rFSH up to the day before GnRH agonist day. The maximum rFSH dose to continue treatment after the first 7 days is 300 IU but the dose could be adjusted when desired.
  As soon as three follicles of 17mm are observed by USS at least, a GnRH agonist (Triptorelin 0.2 mg) will be used for final oocyte maturation at the same day. About 34-36 h thereafter, OPU followed by ICSI is performed. Two days after oocyte pick-up 2 fresh embryos will be transferred
  Arms: ICSI

SUMMARY:
In polycystic ovary syndrome (PCOS) patients, both in vitro maturation (IVM) and intra-cytoplasmic sperm injection (ICSI) are indicated as optional treatments. Although recently ICSI techniques have been reported as more successful the IVM in achieving pregnancy, they have also become much more expensive for the couples involved. Whilst most high-income countries offer Assisted Reproductive Technology (ART) procedures fully or partially paid by the government, the patients in low or middle-income countries have to cover self-fund infertility treatments. With limited resource, a study conducting based on the prevalence - based cost - effectiveness analysis is necessary for health managers, policy makers and especially to assist patients' decision making in these countries.

However, there are still limited published studies that have evaluated the cost-effectiveness of these strategies are available in the literature. This study is conducted based on the prevalence - based cost - effectiveness analysis from the patient's perspective. Activity - based costing method is used to cost in all levels of the healthcare system, which the patients have to pay directly or indirectly. It also analyses incremental cost - effectiveness to evaluate the cost - effectiveness of IVM and ICSI in PCOS women.

DETAILED DESCRIPTION:
A Cost - Effectiveness Analysis (CEA) Study:

* To identify, measure, and evaluate the cost of ICSI treatment and IVM treatment in PCOS patients, and the incremental cost of ICSI system implemented in PCOS patients.
* To quantify the effectiveness of ICSI treatment and the IVM through number and proportion of clinical pregnancy, live birth, and incremental effectiveness of the ICSI treatment implemented in PCOS patients.
* To determine the cost - effectiveness of ICSI treatment compared with IVM in PCOS patients.
* To measure the incremental cost - effectiveness of ICSI treatment implemented. The sample size for this study of 140 subjects, in both groups, being treated for 1 IVM or ICSI cycle is based upon the cost and the effectiveness (live birth rate).

METHODS Cost - Effectiveness Analysis (CEA) Activity - based costing method is used to cost in all levels of the healthcare system which the patients have to pay directly or indirectly for IVM or ICSI. This study also analyzes incremental cost - effectiveness to evaluate the cost - effectiveness of ICSI treatment implemented in PCOS patients.

Sensitivity analysis In this study, two techniques of sensitivity analysis below employing for the decision tree model, which is mentioned as below, are one - way sensitivity analysis and Probabilistic Sensitivity Analysis (PSA).

One - way sensitivity analysis with Tornado diagram will analyses and Probability sensitivity analysis with Monte Carlo simulation and Scatter plots of the difference in costs respecting with the difference in live birth gained will analyses if all parameters varying together simultaneously.

This study also provided the cost - effectiveness acceptability curve (CEAC). The CEAC is applying on the probability sensitivity analysis result, basing on the willingness to pay (WTP). This technique assesses the probability of being cost effective of ICSI treatment comparing to the IVM treatment, respecting to the WTP.

Study Setting: My Duc Hospital Type of data: This study uses a retrospective secondary data collection.

Interventions:

IVM:

* Day 2-4: Ultrasound for Antral Follicles Counts (AFC).
* FSH injection: Day 9, 10 and 11 (can be adjusted 1-3 days before or after to avoid Ultrasound and OPU on holidays). Dose: normally 100 IU/day (maybe 75 - 150 IU/day).
* Follicle and endometrium can be evaluated: on the day of final injection or one day later.
* Cancel this cycle, if pregnancy is detected or suspected ovulation through ultrasound.
* hCG 10.000 IU: one day after the final FSH injection, at 9 p.m. Can be adjusted HCG injection day (± 1-2 days) to avoid Ultrasound and OPU on vacation.
* OPU: 1,5 day after hCG injection (normally 36-42 hours later).
* Sperm collection: on OPU day (if mature follicle presents) or 1 day after OPU day.
* Embryo transfer: 3 days after OPU.
* Luteal support: progesterone gel (90 mg once daily) intra-vaginally and estradiol (4 mg/day PO, twice daily) initiated on the day of OPU or the day thereafter.

ICSI:

Daily SC injections with rFSH - recombinant follicle stimulating hormone (minimum starting dose is around 150 IUI) are started on On day 2 or day 3 of the menstrual cycle (Stimulation Day 1) and continue up to and including Stimulation Day 7.

From Stimulation Day 8 onwards, subjects from ICSI treatment groups will continue with a daily SC dose of rFSH up to the day before Gonadotrophin-releasing hormone (GnRH) agonist day. The maximum rFSH dose to continue treatment after the first 7 days is 300 IU but the dose could be adjusted when desired.

To prevent premature luteinizing hormone (LH) surges the GnRH antagonist (ganirelix acetate SC 0.25 mg/ 0.5 mL) is administered starting on stimulation day 5.

If no follicles ≥ 11mm is visible on the USS on Stimulation day 8, or if no embryo transfer the cycle is to be cancelled. If the ovarian response too high or if there is a risk for Ovarian hyperstimulation syndrome (OHSS), (more than 30 follicles ≥ 11mm on USS), rec-hCG is required to be withheld, and the treatment cycle is to be cancelled.

As soon as three follicles of 17mm are observed by USS at least, a GnRH agonist (Triptorelin 0.2 mg) will be used for final oocyte maturation at the same day. About 34-36 h thereafter, OPU followed by ICSI is performed. Two days after oocyte pick-up 2 fresh embryos will be transferred. Patients with high progesterone level on the trigger day (progesterone level > 2ng/ml), freeze all will be recommended.

Patients using GnRH agonist will have fresh transfer with intense luteal phase support of E2 and P4 (receive intense luteal phase support with E2 and P4 as the same dose mentioned above and progesterone 50 mg i.m. /day), unless patients have high progesterone level on day of trigger (progesterone level > 2ng/ml), freeze all will be recommended.

Frozen embryo transfer cycles:

* Time of starting:

  * Day 2-4 of the cycle.
  * When starting to use drugs, endometrial thickness ≤ 9mm.
* Drugs

  * Estradiol valerate (Valiera 2mg, Progynova 2mg).
  * Starting dose: 8mg/day (Valiera 2mg per os, four times, daily) for 6 days.
* Adjusting dose:

  * Increasing to 12mg/day (Valiera 2mg per os, three times per day, every time 02 tablets) for 5 days if EM thickness < 10mm after 6 days using 8mg/day.
  * Increasing to 16 mg/day (Valiera 2mg per os, four times, every time 2 tablets) for 4 days if EM thickness < 10mm after 5 days using 12mg/day.
  * Attention: Dose up to 16mg/day, patient must be performed ultrasound every 3-4 days for detecting the side effects (headache, dizzy). When this side effect happens, stop your regimen.
  * Maximum treatment interval is 28 days.
* Decide to transfer:

  * Endometrium thickness (EM) ≥ 8mm (this standard doesn't apply to all patients).
  * The minimum time for using estradiol valerate: 10 days.
  * Drug:

    * Progesterone per vagina:

      * Cyclogest 400mg, tid pv, 01 tablet, for 16 days.
      * or Crinone 8% gel, tid pv, 01tube.
    * Estradiol valerate:

      * Valiera 2mg, four times per os, 01 tablet for 16 days.
      * The day for Embryo transfer depends on the age of embryo (Day 2, 3, or 5).

Assessments Before the start of ovarian stimulation, pregnancy is excluded by means of an hCG test, a blood sample is obtained for hormone assessments, and USS is performed to measure and count visible follicles.

Patients will return to the clinic for USS and blood sampling on stimulation days 5 and 8, and the day of hCG or GnRH agonist administration. Additional blood samples will be collected on the day of embryo transfer and 2 weeks after embryo transfer.

Recruitment:

Chief investigator (CI) will review all the medical records and collect all the data (cost, effectiveness, epidemic characteristics...), contacts of PCOS patients. Then CI and colleagues will call the patients for inviting to participate in this project and provide information about the study. If they agree to take part in, collecting data of indirect cost (transportation, administrative costs...) will be provided. The patients have the right to withdraw from the study at any time.

ETHICAL CONSIDERATIONS Institutional Review Board of My Duc Hospital will review the study. The main ethical concerns are whether the research will place the patients at undue risk and whether the subjects are fully informed about the nature of the study. The study will only be conducted after the Ethics Committee approval has been granted.

Ethics approval - From My Duc Hospital Confidentiality - Information sheet de-identified. A unique number is given to each participant. Master list held by CI separately from data.

Declaration of interests - None Access to data - Investigators only Ancillary and post-trial care - None

ELIGIBILITY:
Include:

* Couples undergoing IVM or ICSI treatment for the 1st time.
* Husband: total mobile sperm count over 10 million/ml (before washing) or over 2 million/ml (after washing) or normal semen analysis (WHO 2010 criteria).
* Wife: PCOS patients (Rotterdam European Society of Human Reproduction and Embryology (ESHRE)/ American Society of Reproductive Medicine (ASRM) 2004 aged from 18 to 37 at the time of conducting IVM or ICSI.
* Each subject must have results of clinical laboratory test (complete blood count (CBC), blood chemistries, and urinalysis, pap smear) within normal limits or clinically acceptable to the investigator, as measured by the local laboratory at screening.
* Each subject must have results of a physical examination, including blood pressure, within normal limits or clinically acceptable limits to the investigator.

Exclude:

* The subject (wife) has a recent (i.e. within 3 years prior to conducting IVM or ICSI) history of/ or any current endocrine abnormality (irrespective whether the patient is stabilized on treatment).
* The subject has a recent history of/or current epilepsy, thrombophilia, diabetes, cardiovascular, gastro-intestinal, hepatic, renal or pulmonary or auto-immune disease requiring regular treatment.
* Endometriosis (in uterine muscle, ovary or pelvis) or IVF/ICSI with donated sperm, donated eggs or IVM with donated sperm, clomiphene citrate resistant PCOS (PCOS), tubal factor (blocked fallopian tube, hydrosalpinx), abnormal uterine structure (submucosal fibroid or intramural fibroid ≥30 mm, uterine polyp, bicornuate uterus, didelphic uterus).
* The subject has tested positive for Human Immunodeficiency Virus (HIV) or Hepatitis B (by the local laboratory; results obtained within one year prior to conducting IVM or ICSI are considered valid).
* The subject has contraindications for the use of gonadotropins (ex; tumors, pregnancy/lactation, undiagnosed vaginal bleeding, hypersensitivity, or ovarian cysts) or GnRH-antagonist (e.g. hypersensitivity, pregnancy/lactation).
* The subject has known gene defects, genetic abnormalities, or abnormal karyotyping, relevant for the current indications or for the health of the offspring.
* The subject smokes or has recently stopped smoking (ex. within the last 3 months).
* The subject has a history or presence of alcohol or drug abuse within 12 months prior to conduct IVM or ICSI.
* The subject has used any experimental drugs within 3 months prior to conduct IVM or ICSI.
* The subject is participating in any other clinical study (excluding surveys).
* Those who do not complete the process of IVM or IVF/ICSI (withdrawing, no embryo for transfer or embryos haven't been transferred).

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
live birth | 36 weeks
  the complete expulsion or extraction from its mother of a product of conception, irrespective of the duration of the pregnancy, which, after such separation, breathes or shows any other evidence of life - e.g. beating of the heart, pulsation of the umbilical cord or definite movement of voluntary muscles - whether or not the umbilical cord has been cut or the placenta is attached. Each product of such a birth is considered live born (WHO).
direct costs | 1 year
  the costs (Vietnam dong) for medical services, medication, examinations, procedures, etc.
indirect costs | 1 year
  the costs (Vietnam dong) for patients' working hour loss (income per one working hour x number of hours), transportation fee (by motorbike, car, bus, taxi, others), accommodation (including hotel, guest house, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Khoa D Le, Dr, Principal Investigator — Mỹ Đức Hospital

IPD SHARING:
Plan to Share IPD: No